CLINICAL TRIAL: NCT04629352
Title: Examining Neuroplasticity Modulation as Mechanistic Basis of tDCS Treatment Effects on Auditory Verbal Hallucination in Schizophrenia
Brief Title: Effect of Neuroplasticity Modulation in tDCS Treatment Response Among Schizophrenia Patients With Auditory Hallucination
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Anushree Bose, Principal Investigator, National Institute of Mental Health and Neuro Sciences, India
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IA/CPHE/19/1/504591
Record Dates: First submitted 2020-11-02; First posted 2020-11-16 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Auditory verbal hallucination; Transcranial Direct Current stimulation (tDCS); Schizophrenia; Neuroplasticity; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hallucinations

STUDY DESIGN:
Intervention Model Description: This prospective longitudinal study will administer add-on accelerated tDCS to SCZ patients in a double-blind, randomised, parallel-arm sham-controlled design. In the accelerated tDCS protocol, 10 sessions (5 sessions per day) will be administered over 2 days. Patients who show ≥20% reduction in AVH severity will be followed up at one month and three months after completion of tDCS-RCT, and other patients will be offered clinician-determined treatment, including open-label accelerated tDCS treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A computer-generated randomization sequence will be used for random assignment of treatment condition. A tDCS device equipped to deliver verum or sham stimulation upon entering manufacturer-assigned codes will be used for the study. Allocation concealment will be maintained by off-site bio-statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Verum Accelerated Transcranial Direct Current Stimulation (acctDCS) (Experimental): Each SCZ patient will receive five sessions daily for two days, a 10-session course of tDCS [anode: left-DLPFC (at F3) and cathode: left-TPJ (midway between C3 and P3); electrode size: 35cm2]. For the Verum-tDCS condition, 2-mA of constant current will be delivered for 20 minutes, with additional ramp-up and ramp-down of 30 seconds each.
  Interventions: Device: Verum Accelerated Transcranial Direct Current Stimulation (acctDCS)
- Sham Accelerated Transcranial Direct Current Stimulation (tDCS) (Placebo Comparator): Each SCZ patient will receive five sessions daily for two days, a 10-session course of tDCS [anode: left-DLPFC (at F3) and cathode: left-TPJ (midway between C3 and P3); electrode size: 35cm2]. For Sham-tDCS, no current will be delivered beyond the initial ramp-up time.
  Interventions: Device: Sham Accelerated Transcranial Direct Current Stimulation (acctDCS)

INTERVENTIONS:
Device: Verum Accelerated Transcranial Direct Current Stimulation (acctDCS) — In verum transcranial direct current stimulation (tDCS), patient will receive five sessions daily for two days, a 10-session course of tDCS [anode: left-DLPFC (at F3) and cathode: left-TPJ (midway between C3 and P3); electrode size: 35cm2]. For Verum-tDCS condition, 2-mA of constant current will be delivered for 20-minutes, additional ramp-up and ramp-down of 20 seconds each.
  Arms: Verum Accelerated Transcranial Direct Current Stimulation (acctDCS)
Device: Sham Accelerated Transcranial Direct Current Stimulation (acctDCS) — In sham transcranial direct current stimulation (tDCS), each SCZ patient will receive five sessions daily for two days, a 10-session course of tDCS [anode: left-DLPFC (at F3) and cathode: left-TPJ (midway between C3 and P3); electrode size: 35cm2]. However, no current will be delivered beyond initial ramp-up time though the tDCS device display will indicate that 2mA current is being applied.
  Arms: Sham Accelerated Transcranial Direct Current Stimulation (tDCS)

SUMMARY:
Schizophrenia is a severe neuropsychiatric disorder of the brain and is also one of the top ten disabling diseases. A common symptom of schizophrenia (SCZ) is hearing voices inside one's heads which others do not. Despite adequate medication, SCZ patients may continue to hear voices that are often rude or unfriendly and cause distress to the patients. Transcranial direct current stimulation (tDCS) is a safe, non-invasive brain stimulation technique that reduces 'hearing voices'. However, how and why add-on tDCS works is unclear. The brain can change itself in response to its environment; this is called neuroplasticity. tDCS possibly changes the brain's environment and/or enhances the brain's ability to respond favourably to its environment. This theory will be examined here by studying changes in brain functions before and after giving tDCS to schizophrenia patients hearing voices. The aim of this study is to examine the brain's neuroplasticity potential as the biological phenomena driving treatment effects of tDCS in Schizophrenia patients with clinically significant and persistent auditory verbal hallucinations. The secondary aims are to answer whether the brain's neuroplasticity potential in schizophrenia patients can predict their responsivity to tDCS treatment for auditory verbal hallucinations, and if chronicity of illness effects tDCS treatment response.

The brain's neuroplasticity potential will be examined using neuroimaging and neurophysiological techniques that give information about the integrity of the brain's signal processing efficiency, the chemical concentration of certain bio-molecules within it, and how well different areas of the brain communicate with each other. With this information, the potential role of the brain's neuroplasticity potential in facilitating treatment effects of tDCS can be better understood. With this knowledge, it could be possible personalize tDCS treatment, profile tDCS responders and non-responders based on demographic and biological factors, and prescribe tDCS at the appropriate time within the illness course for maximal benefit to the SCZ patients.

DETAILED DESCRIPTION:
20-30% schizophrenia (SCZ) patients struggle with auditory verbal hallucinations (AVH) minimally responsive to pharmaceutical treatments. An add-on fronto-temporoparietal transcranial direct current stimulation (tDCS) is suggested to address persistent AVH in SCZ patients. High heterogeneity among existing randomized control trials for AVH treatment in SCZ and the lack of empirical studies investigating the tDCS action mechanism warrants a systematic investigation into the mechanistic basis of tDCS action.

This proposal aims to examine the potential for neuroplasticity modulation as the mechanistic factor behind the therapeutic effects of left fronto-temporo-parietal tDCS for treating clinically significant AVH in early-course and chronic SCZ patients. It has been proposed and demonstrated that more tDCS sessions over a shorter interval lead to rapid plasticity induction. Accelerated tDCS protocol delivers a higher number of tDCS sessions over a shorter duration. Accelerated protocol (5 sessions/day for 2 days, inter-session interval~20 minutes) for the treatment of AVH in SZ showed clinical improvement with concurrent changes in neurophysiological correlates of auditory hallucination pathophysiology. Specifically, this study will examine neuroplasticity potential as a biomarker for tDCS treatment response with an accelerated tDCS (acctDCS) protocol. Using a randomized, double-blind, sham-controlled parallel-arm, pre-post design, changes in neuroplasticity potential with tDCS treatment for AVH in SCZ will be assessed. The four composite primary outcome measures of this study are:

1. changes in N100-derived event-related-potential waveforms (neurophysiological),
2. changes glutamine-glutamate levels (neurochemical),
3. changes in resting-state functional connectivity (neuroimaging), and
4. reduction in AVH severity (clinical).

The secondary objectives of this study are:

1. exploring the correlation between neurobiological measures of neuroplasticity changes induced by tDCS and clinical improvement in AVH to indicate the nature and strength of the relationship between the two;
2. exploring the effect of verum (active) tDCS on early course versus late course SCZ patients will uncover if illness chronicity is a potential barrier to tDCS responsivity; and
3. utilizing disorder-related (age at illness onset, medication, the severity of the symptom, etc.) and biographic (age, sex, years of education, etc.) features of the study sample towards predicting neuroplasticity modulation in the study sample.

ELIGIBILITY:
INCLUSION CRITERIA

* Diagnosis of schizophrenia or schizoaffective disorder as per DSM-5 (American Psychiatric Association, 2013)
* Clinically Significant Auditory Verbal Hallucinations
* Right-handedness
* Written informed consent

EXCLUSION CRITERIA

* Features suggestive of a psychiatric emergency
* Any contraindication to tDCS procedures
* Pregnancy or post-partum status
* Left/Mixed Handedness

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Neurophysiological Measure: Change in amplitude of N100-related waveforms | Baseline: Day-1, After single session of tDCS: Day-1, Day-6: After 10 sessions of RCT tDCS
  Event-related potential (N100) based indices of changes in early auditory processing and adaptive plasticity in response to tDCS treatment.
Neuro-Chemical Measure: Change in concentration of glutamate-glutamine levels | Baseline: Day-1, Day-6: After 10 sessions of RCT tDCS
  Spectroscopy based indices of glutamate-glutamine levels at left temporo-parietal junction (TPJ) and left prefrontal cortex (PFC) in response to tDCS treatment.
Neuro-haemodynamic Measure: Change in strength of resting-state-functional-connectivity among brain areas | Baseline: Day-1, Day-6: After 10 sessions of RCT tDCS
  Neuroimaging based indices of seed-based resting-state-functional-connectivity (rs-FC) of the left-TPJ with left-PFC in response to tDCS treatment.
Clinical Measure: Change in auditory verbal hallucination score | Baseline: Day-1, Day-6: After 10 sessions of RCT tDCS, One month Follow-up, Three-months follow-up
  Change in auditory hallucination severity as indicated by Auditory Hallucination Rating Scale (AHRS) scores. Minimum score is 2 and maximum score is 41. Higher the score more severe the symptom.

SECONDARY OUTCOMES:
Change in auditory hallucination severity in responsive schizophrenia patients (with ≥25% reduction in auditory hallucination severity at post RCT time point) at 1-month and 3-month follow-up | One-month Follow-up, Three-month follow-up
  Change in auditory hallucination severity as indicated by Auditory Hallucination Rating Scale at (AHRS) scores at clinical follow-up. Minimum score is 2 and maximum score is 41. Higher the score more severe the symptom.
Change in auditory hallucination score in early course and late course schizophrenia patients | Baseline: Day-1, Day-6: After 10 sessions of RCT tDCS
  Both Early course (illness duration ≤2 years; n=36) and Late course (illness duration ≥5 years; n=36) schizophrenia patients will be recruited to explore the influence of illness chronicity on neuroplasticity potential and tDCS responsivity. Change in auditory hallucination severity as indicated by Auditory Hallucination Rating Scale at (AHRS) scores. Minimum score is 2 and maximum score is 41. Higher the score more severe the symptom.

OTHER OUTCOMES:
In a posthoc analysis, a prediction model for the potential of neuroplasticity modulation with tDCS will be attempted using machine learning algorithms and Bayesian approaches. | Day-6: After 10 sessions of RCT tDCS, One-month follow-up
  Disorder-related (age at illness onset, medication, severity of symptom, etc.) and biographic features (age, sex, years of education, etc.) of the study sample will be used to develop a prediction model for neuroplasticity modulation in this study sample. This model will be optimized further at one-month to take into account the changes in auditory verbal hallucination severity at follow-up among SCZ patients responsive to tDCS.

CONTACTS AND LOCATIONS:
Overall Officials: Anushree Bose, PhD, Principal Investigator — Department of Psychiatry, NIMHANS, Bengaluru, Karnataka, India; Ganesan Venkatasubramanian, MD, PhD, Study Chair — Professor at Department of Psychiatry, NIMHANS, Bengaluru, Karnataka, India
Locations (1):
- Department of Psychiatry, National Institute of Mental Health And Neuro Sciences (NIMHANS), Bengaluru, Karnataka, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
De-identiﬁed individual participant data (IPD) that underlie the results reported in specific publication arising out of the trial will be shared with researchers for individual participant data meta-analysis.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD will be shared 9 months after the publication of the trial results and will stay available for up to 36 months.
Access Criteria: Researchers seeking to access IPD should write to the investigator(s) with a methodologically sound proposal. The investigator(s) will provide the details of further steps.